CLINICAL TRIAL: NCT02464384
Title: Multicenter, Prospective, Open-label, Cohort Study With Collection of Blood Samples and Ultrasound / MRI and X-ray Examination
Brief Title: Prediction of Erosive Disease in Early Rheumatoid Arthritis (RA) by Ultrasound and Cartilage Biodegradation Markers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPEDRA01_01.07.2013
Record Dates: First submitted 2015-02-10; First posted 2015-06-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Erosive Disease in Early Rheumatoid Arthritis
Keywords: ultrasound and cartilage biodegradation markers
MeSH Terms: interventions — Phlebotomy; High-Energy Shock Waves; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cohort study (Other): Collection of blood samples and ultrasound / MRI and x-ray examination.
  Interventions: Procedure: Venipuncture, ultrasound, MRI, x-ray

INTERVENTIONS:
Procedure: Venipuncture, ultrasound, MRI, x-ray — Collection of blood samples and ultrasound / MRI and x-ray examination

SUMMARY:
Multicenter, prospective, open-label, cohort study. Primary objective: Determination of the predictive value of US alone and in combination with cartilage biodegradation markers on radiographic progression (change in Ratingen score)

Secondary objectives:

* Correlation of ultrasound synovitis score and clinical disease activity score
* Determination of the sensitivity of ultrasound erosion detection compared to MRI
* Assessment of the value of including tenosynovitis assessment for predicting radiographic progression
* Assessment of the predictive value of ultrasound synovitis score at baseline for the need to install biologic DMARDs

DETAILED DESCRIPTION:
Multicenter, prospective, open-label, cohort study with collection of blood samples and ultrasound / MRI and x-ray examination.

Duration of study: 12 months This study is a prospective cohort study. The choice of therapy at any time during the study is entirely up to the treating rheumatologist. The study does not put any restriction on the management of the patient which will be according to routine care.

At occurrence of one or more of the above mentioned variables defining adverse clinical outcome (prednisone in a dose exceeding 10mg/d and/or intraarticular steroid injections and/or start of biologic DMARD) an analysis as for D360 will be performed US-Score: SONAR-Score assessment of synovitis (22 joints)/erosions (14 joints)/cartilage thickness (8 joints) Clinical evaluation: Disease activity score (DAS28 = Number of tender and swollen joints (0-28), additional measures (ESR / CRP), Patient Global Health (0-100), health assessment questionnaire (HAQ) at 0, 3, 6, 9, 12 months (attached) Lab: ESR, CRP Serology: Antinuclear antibody (ANA), Rheumatoid factor (RF), Anti-cyclic citrullinated peptide (anti-CCP) at baseline if not available COL2-1 / COL2-1N X-Ray: hands and feet at baseline and 12 months (scoring according to Ratingen Score) if not available MRI without contrast at baseline and at 12 months or when first erosions detected with US

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling all of the following inclusion criteria may be enrolled in the study:
* male and female subjects, Age above 18 yrs
* recent onset RA fulfilling the American College of Rheumatology (ACR) criteria (revised 2010)
* Symptoms for at least 6 weeks
* no previous DMARD treatment
* no intraarticular steroid injections in the last 4 weeks before inclusion
* no treatment with oral steroids exceeding the equivalent of 10mg prednisone per day in the last 2 weeks before inclusion
* signed Informed Consent after being informed

Exclusion Criteria:

* History of inflammatory joint disease other than RA
* History of active Tbc, histoplasmosis or listeriosis
* History of lymphoma or other malignancies within 5 years
* Contraindication for the use of DMARD's or biologics
* Comorbidities: severe myocardial dysfunction, recent stroke (within 3 months), uncontrolled diabetes and other disease which in the opinion of the investigator, would put the subject at risk by participation in the trial
* History of demyelinating disorders
* persistent or recurrent infections
* Pregnancy or breast feeding
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Determination of the predictive value of US alone and in combination with cartilage biodegradation markers on radiographic progression (change in Ratingen score) | 12 months

SECONDARY OUTCOMES:
Correlation of ultrasound synovitis score and clinical disease activity score | 12 months
Determination of the sensitivity of ultrasound erosion detection compared to MRI | 12 months
Assessment of the value of including tenosynovitis assessment for predicting radiographic progression | 12 months
Assessment of the predictive value of ultrasound synovitis score at baseline for the need to install biologic DMARDs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ciurea, MD, Principal Investigator — Department of Rheumatology, University Hospital Zurich